CLINICAL TRIAL: NCT05312879
Title: A Phase 2/3 Adaptive, Double-blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of VX-147 in Adult and Pediatric Subjects With APOL1-mediated Proteinuric Kidney Disease
Brief Title: Phase 2/3 Adaptive Study of VX-147 in Adult and Pediatric Participants With APOL1- Mediated Proteinuric Kidney Disease
Acronym: AMPLITUDE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX21-147-301; 2024-515633-15-00 (Other: EU Trial (CTIS) Number)
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-08

CONDITIONS: Proteinuric Kidney Disease
Keywords: APOL1-mediated kidney disease (AMKD)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 2: VX-147 (Experimental): Participants will be randomized to receive different dose levels of VX-147.
  Interventions: Drug: VX-147
- Phase 2: Placebo (Placebo Comparator): Participants will receive placebo matched to VX-147.
  Interventions: Drug: Placebo
- Phase 3: VX-147 (Experimental): Participants will receive VX-147 with the dose to be based on the outcome of Phase 2.
  Interventions: Drug: VX-147
- Phase 3: Placebo (Placebo Comparator): Participants will receive placebo matched to VX-147.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX-147 — Tablets for oral administration.
  Arms: Phase 2: VX-147; Phase 3: VX-147
Drug: Placebo — Tablets for oral administration.
  Arms: Phase 2: Placebo; Phase 3: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, tolerability, and pharmacokinetics (PK) of VX-147 in adult and pediatric participants with apolipoprotein L1 (APOL1)-mediated proteinuric kidney disease.

ELIGIBILITY:
Key Inclusion Criteria:

* APOL1 genotype of G1/G1, G2/G2, or G1/G2
* Proteinuric kidney disease

Key Exclusion Criteria:

* Solid organ or bone marrow transplant
* Uncontrolled hypertension
* History of diabetes mellitus
* Known underlying cause of kidney disease including but not limited to sickle cell disease

Other protocol defined Inclusion/Exclusion criteria apply.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 466 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in Urine Protein to Creatinine Ratio (UPCR) at Week 48 (Assessed at the Week 48 Interim Analysis) | From Baseline at Week 48
Estimated Glomerular Filtration Rate (eGFR) Slope Assessed at the Week 48 Interim Analysis | From Baseline Through >= Week 48
eGFR Slope Assessed at Study Completion | From Baseline Through Study Completion (Approximately 2 Years After the Last Participant Enrolls)

SECONDARY OUTCOMES:
Time to Composite Clinical Outcome of a Sustained Decline of >=30 Percent (%) in eGFR, the Onset of end-stage Kidney Disease or Death | From Baseline Through Study Completion (Approximately 2 Years After the Last Participant Enrolls)
Safety and Tolerability as Assessed by Number of Participants With Adverse events (AEs) and Serious Adverse Events (SAEs) | Day 1 Through Study Completion (Approximately 2 Years After the Last Participant Enrolls)
Maximum Plasma Concentration (Cmax) of VX-147 | Day 1 and Week 40
Area Under the Concentration Versus Time Curve During a Dosing Interval (AUCtau) of VX-147 | Day 1 and Week 40
Observed Pre-dose Plasma Concentration (Ctrough) of VX-147 | Day 1 up to Week 40
Acceptability Tablet Formulation of VX-147 in Pediatric Participants using the Convenience Domain of the Treatment Satisfaction Questionnaire for Medication (TSQM) Version 1.4 | Day 1 and Week 48

CONTACTS AND LOCATIONS:
Locations (318):
- United States (227):
  - Alabama Kidney Research, Alabaster, Alabama
  - EmVenio Research - Mobile Unit - Birmingham, Birmingham, Alabama
  - Cardiology, P.C., Birmingham, Alabama
  - Children's Hospital of Alabama, Birmingham, Alabama
  - The Kirklin Clinic - Nephrology, Birmingham, Alabama
  - Nephrology Associates, Fairhope, Alabama
  - Heart Center Research LLC, Huntsville, Alabama
  - Nephrology Consultants, LLC, Huntsville, Alabama
  - Renal Associates of Alabama, LLC, Montgomery, Alabama
  - Arizona Kidney Disease and Hypertension Center - Banner Desert Office, Mesa, Arizona
  - Arizona Kidney Disease and Hypertension Center - Thomas Office, Phoenix, Arizona
  - Phoenix Children's Hospital, Inc. - Nephrology, Phoenix, Arizona
  - CHI St. Vincent Heart Clinic Arkansas- Cardiology and Medicine Clinic - Little Rock, Little Rock, Arkansas
  - UAMS Medical Center - Pulmonology, Little Rock, Arkansas
  - The Medical Research Group - Saint Agnes Medical Center, Fresno, California
  - Amicis Research Center - Balboa, Granada Hills, California
  - Kidney Care Center of North Valley, Granada Hills, California
  - Eastside Clinical Research Associates, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA Division of Nephrology, Los Angeles, California
  - UCI Center for Clinical Research, Orange, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Helen Diller Medical Center at Parnassus Heights, San Francisco, California
  - UCLA Lundquist Institute at Harbor-UCLA Medical Center, Torrance, California
  - Kidney and Hypertension Center, Victorville, California
  - Greater Hartford Nephrology, Bloomfield, Connecticut
  - Nephrology & Hypertension Associates, PC, Middlebury, Connecticut
  - Yale University - Yale Nephrology Clinical Research Clinic, New Haven, Connecticut
  - Children's National Hospital - Nephrology, Washington D.C., District of Columbia
  - The George Washington University - GW Medical Faculty Associates, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington D.C, Washington D.C., District of Columbia
  - Bay Pines Foundation, Bay Pines, Florida
  - Nova Clinical Research, LLC - Bradenton - 59th St, Bradenton, Florida
  - Clinical Research of Brandon, LLC, Brandon, Florida
  - AMR-Miami, Coral Gables, Florida
  - Horizon Research Group - Coral Gables, Coral Gables, Florida
  - South Florida Nephrology Research, Coral Springs, Florida
  - Delray Physician Care Center, Delray Beach, Florida
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - Shands Hospital - Nephrology, Gainesville, Florida
  - Velocity Clinical Research - Hallandale Beach, Hallandale, Florida
  - Qway Research, Hialeah, Florida
  - Elixia Pines, Hollywood, Florida
  - UF Health Cardiovascular Center - Jacksonville, Jacksonville, Florida
  - South Florida Research Institute, Lauderdale Lakes, Florida
  - Total Research Group, LLC, Miami, Florida
  - MedBio Trials, Miami, Florida
  - Cordova Research Institute, Miami, Florida
  - South Florida Research, Miami Springs, Florida
  - CTR Oakwater, LLC, Orlando, Florida
  - Synexus Clinical Research - Orlando, Orlando, Florida
  - Omega Research Orlando, LLC - Mercy Dr, Orlando, Florida
  - Infigo Clinical Research, Sanford, Florida
  - Genesis Clinical Research, Tampa, Florida
  - Elixia Tampa, Tampa, Florida
  - American Clinical Trials LLC - Acworth, Acworth, Georgia
  - Kaiser Permanente Georgia, Atlanta, Georgia
  - Emory School of Medicine - Renal Division, Atlanta, Georgia
  - Advanced Clinical Research of Atlanta, Atlanta, Georgia
  - Morehouse School of Medicine, Grady Memorial Hospital, Atlanta, Georgia
  - Emory Childrens Center - Nephrology, Atlanta, Georgia
  - Synexus Clinical Research - Atlanta (DRS), Atlanta, Georgia
  - Fides Clinical Research, Atlanta, Georgia
  - Augusta University Medical College of Georgia - Adult Sickle Cell Clinic, Augusta, Georgia
  - Coastal Medical Research, Brunswick, Georgia
  - Randomize Now - College Park, College Park, Georgia
  - Clincept - Veterans Pkwy., Columbus, Georgia
  - Renal Associates, Columbus, Georgia
  - Georgia Nephrology - Decatur, Decatur, Georgia
  - Atlanta VA Healthcare System, Decatur, Georgia
  - American Clinical Trials LLC - Douglasville, Douglasville, Georgia
  - Southeast Kidney Associates, East Point, Georgia
  - Javara Inc./Privia Medical Group - Fayetteville, GA, Fayetteville, Georgia
  - Georgia Nephrology - Lawrenceville - Billing Office, Lawrenceville, Georgia
  - Javara Inc./Privia Medical Group - Savannah, GA, Savannah, Georgia
  - Inova Clinical Trials and Research Center, Tyrone, Georgia
  - Rophe Adult and Pediatric Medicine, Union City, Georgia
  - Synexus Clinical Research - Chicago (DRS), Chicago, Illinois
  - EmVenio Research - Chicago, Chicago, Illinois
  - Ann & Robert H. Lurie Children's Hospital of Chicago - Nephrology, Chicago, Illinois
  - Northwestern Medical Group, Chicago, Illinois
  - UChicago Medicine - Comer Children's Hospital, Chicago, Illinois
  - NANI Research LLC - Evergreen Park IL, Evergreen Park, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Essential Concepts Research Solutions, Palos Hills, Illinois
  - NANI Research LLC - Fort Wayne IN, Fort Wayne, Indiana
  - IU School of Medicine - Nephrology, Indianapolis, Indiana
  - Nephrology Physicians, LLC, Mishawaka, Indiana
  - University of Iowa Health Care Medical Center- Nephrology, Iowa City, Iowa
  - Clinical & Translational Science Unit (CTSU) - Nephrology, Kansas City, Kansas
  - Premier Clinical Research, Overland Park, Kansas
  - Renal Associates of Baton Rouge, Baton Rouge, Louisiana
  - LCMC Health, Metairie, Louisiana
  - Barnum Medical Research - Bienville St, Natchitoches, Louisiana
  - Louisiana Clinical and Translational Science (LA CaTS) Center, New Orleans, Louisiana
  - University Medical Center - New Orleans - Nephrology, New Orleans, Louisiana
  - Ochsner Medical Center - New Orleans, New Orleans, Louisiana
  - Northwest Louisiana Nephrology, LLC, Shreveport, Louisiana
  - Louisiana State University Health Shreveport, Shreveport, Louisiana
  - Monroe Research, LLC, West Monroe, Louisiana
  - Javara Inc./Privia Medical Group - Annapolis, MD, Annapolis, Maryland
  - University of Maryland Medical Center - General Clinical Research Center, Baltimore, Maryland
  - The Johns Hopkins University - Johns Hopkins Hospital - Nephrology, Baltimore, Maryland
  - Mid-Atlantic Permanente Research Institute, Gaithersburg, Maryland
  - Patient First Clinical Trials, Lutherville, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Javara Inc./Privia Medical Group - Silver Spring, MD - Columbia Pike, Silver Spring, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center - Nephrology, Boston, Massachusetts
  - Whittier Street Health Center, Roxbury, Massachusetts
  - Renal and Transplant Associates of New England, PC, Springfield, Massachusetts
  - Kidney Care and Transplant Services of New England - West Springfield, West Springfield, Massachusetts
  - A. Alfred Taubman Health Care Center - Nephrology Clinic at Taubman Center, Ann Arbor, Michigan
  - Henry Ford Health System - Nephrology, Detroit, Michigan
  - Quest Research Institute, Farmington Hills, Michigan
  - AA Medical Research Center, Flint, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - St. Clair Nephrology Research, Roseville, Michigan
  - Center for Advanced Kidney Research, Saint Clair Shores, Michigan
  - InterMed Consultants - Edina Clinic, Edina, Minnesota
  - Minneapolis VA Healthcare System, Minneapolis, Minnesota
  - Nephrology Associates, P.C. - Columbus, Columbus, Mississippi
  - Prime Health and Wellness, Fayette, Mississippi
  - UMMC Grenada Hospital, Grenada, Mississippi
  - G.V. (Sonny) Montgomery VAMC, Jackson, Mississippi
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - SKY Integrative Medical Center, Ridgeland, Mississippi
  - Nephrology and Hypertension Associates - Tupelo, Tupelo, Mississippi
  - Center for Specialized Medicine - Nephrology, St Louis, Missouri
  - Barnes-Jewish Center for Outpatient Health, St Louis, Missouri
  - St. Louis Children's Hospital - Nephrology, St Louis, Missouri
  - St. Louis Heart and Vascular, P.C., St Louis, Missouri
  - Nevada Kidney Disease and Hypertension Centers, Las Vegas, Nevada
  - DaVita Kidney Care - Las Vegas, Las Vegas, Nevada
  - CUH - Sheridan Pavilion - Three Cooper Plaza, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Bioluminux Clinical Research New Jersey, Hamilton, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Rutgers Doctors Office Center, Newark, New Jersey
  - New Mexico VA Healthcare System, Albuquerque, New Mexico
  - Renal Medicine Associates, Albuquerque, New Mexico
  - Kings County Hospital, Brooklyn, New York
  - SUNY Downstate Health Sciences University, Brooklyn, New York
  - Clindove Research LLC, Brooklyn, New York
  - New York Presbyterian Queens, Flushing, New York
  - Zucker School of Medicine, Great Neck, New York
  - Scott Research, Inc., Laurelton, New York
  - VA New York Harbor Healthcare System, New York, New York
  - Grossman School of Medicine, New York, New York
  - Synexus Clinical Research - New York (DRS), New York, New York
  - The Rogosin Kidney Center, New York, New York
  - Icahn School of Medicine at Mount Sinai - Nephrology, New York, New York
  - General Nephrology Clinic - New York City, New York, New York
  - NYC Health + Hospital/Harlem, New York, New York
  - Kidney Medical Associates, PLLC, The Bronx, New York
  - Montefiore Einstein - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Einstein Hospital - Moses Campus, The Bronx, New York
  - James J. Peters VA Medical Center, The Bronx, New York
  - North Carolina Nephrology P.A. - Cary, Cary, North Carolina
  - UNC Clinical and Translational Research Center, Chapel Hill, North Carolina
  - Metrolina Nephrology Associates - Freedom Dr, Charlotte, North Carolina
  - Duke University Hospital - Children's Health Center, Durham, North Carolina
  - Eastern Nephrology Associates - Greenville Office, Greenville, North Carolina
  - Eastern Nephrology Associates - Jacksonville Office, Jacksonville, North Carolina
  - Eastern Nephrology Associates - Kinston Office, Kinston, North Carolina
  - Eastern Nephrology Associates - New Bern Office, New Bern, North Carolina
  - Eastern Nephrology Associates - Wilmington Office, Wilmington, North Carolina
  - Brookview Hills Research Associates, Winston-Salem, North Carolina
  - UC - DCI McMillan Research Unit, Cincinnati, Ohio
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - Louis Stokes Cleveland VA medical Center, Cleveland, Ohio
  - UH Cleveland Medical Center - Nephrology, Cleveland, Ohio
  - Cleveland Clinic - Main Campus, Cleveland, Ohio
  - Ohio State University - Wexner Medical Center - Nephrology Clinical Trials Unit, Columbus, Ohio
  - Jefferson Health - 33 South 9th Street, Philadelphia, Pennsylvania
  - Lewis Katz School of Medicine at Temple University - Section of Nephrology, Philadelphia, Pennsylvania
  - Jefferson Einstein Philadelphia Hospital - Nephrology, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh - Nephrology, Pittsburgh, Pennsylvania
  - Lifespan Clinical Research Center, East Providence, Rhode Island
  - Pharmacorp Clinical Trials, Inc, Charleston, South Carolina
  - Medical University of South Carolina - Pulmonology, Charleston, South Carolina
  - Columbia Nephrology Associates, PA, Columbia, South Carolina
  - Carolina Nephrology, PA, Spartanburg, South Carolina
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - Le Bonheur Children's Hospital - Outpatient Clinic, Memphis, Tennessee
  - CNS Healthcare - Memphis, Memphis, Tennessee
  - Nashville General Hospital - Meharry Medical College - Nephrology, Nashville, Tennessee
  - Nashville VA Medical Center, Nashville, Tennessee
  - Nephrology Clinical Trials Center, Nashville, Tennessee
  - Dallas Renal Group - Mansfield, Arlington, Texas
  - Arlington Nephrology, Arlington, Texas
  - Baylor Scott and White Research Institute - Nephrology, Dallas, Texas
  - Dallas Renal Group- Dallas, Dallas, Texas
  - Zenos Clinical Research, Dallas, Texas
  - Nephrotex Research Group, Dallas, Texas
  - Dallas Renal Group - Liberty Dallas Dialysis Center, Dallas, Texas
  - Dallas Nephrology Associates - Dallas Landry Office, Dallas, Texas
  - Southwest Family Medicine Associates (SFMA) - Dallas, Dallas, Texas
  - UTSW Medical Center - Nephrology, Dallas, Texas
  - Davita Clinical Research - El Paso, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Prolato Clinical Research Center - Kirby Dr, Houston, Texas
  - Ronald Ralph MD PA, Houston, Texas
  - Houston Medical Research Institute, LLC, Houston, Texas
  - Clinical Research Strategies - Romano North Main Office, Houston, Texas
  - Frenova-Southwest Houston, Houston, Texas
  - NTKDA Lewisville, Lewisville, Texas
  - Prime Clinical Research Inc - Lewisville, Lewisville, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Prime Clinical Research - Mansfield - Regency Parkway, Mansfield, Texas
  - San Antonio Kidney Disease Center Physicians Group - Medical Center, San Antonio, Texas
  - University of Texas Health Science Center - Nephrology, San Antonio, Texas
  - San Antonio Kidney Disease Center Physicians Group - Westover Hills, San Antonio, Texas
  - Kidney Specialists of N Houston, PLLC, Shenandoah, Texas
  - Renal Research of Montgomery County, PLLC, The Woodlands, Texas
  - Tranquil Clinical Research, Webster, Texas
  - UVA Health - Nephrology Clinical Research Center, Charlottesville, Virginia
  - Tidewater Kidney Specialists - Church St., Norfolk, Virginia
  - York Clinical Research, LLC, Norfolk, Virginia
  - McGuire Research Institute, Inc. (151), Richmond, Virginia
  - Virginia Commonwealth University - Division of Nephrology, Richmond, Virginia
  - Nephrology Associates of Tidewater, LTD, Virginia Beach, Virginia
  - UW Medical Center - Montlake - Nephrology, Seattle, Washington
  - Medical College of Wisconsin - Pulmonology, Milwaukee, Wisconsin
  - Milwaukee Nephrologists - Wauwatosa, Wauwatosa, Wisconsin
- Belgium (2):
  - Universite Catholique de Louvain - Pulmonology, Woluwe-Saint-Lambert, Brussels Capital
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg - Pulmonology, Leuven
- Brazil (29):
  - Centro de Pesquisa Clinica do Coracao, Aracaju
  - Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte
  - Faculdade de Medicina de Botucatu - CKD and Hypertension Department, Botucatu
  - Faculdade de Medicina de Botucatu - Kidney Transplantation Department, Botucatu
  - IPECC - Instituto de Pesquisa Clinica de Campinas, Campinas
  - Instituto Pro-Renal, Curitiba
  - PUC Trials - Unidade Epicenter, Curitiba
  - Instituto de Ensino e Pesquisa Clinica do Ceara, Fortaleza
  - Walter Cantídio University Hospital, Fortaleza
  - Federal University of Goiás (UFG), Goiânia
  - Cmip-Centro Mineiro de Pesquisa Ltda, Juiz de Fora
  - Galileo Medical Research Ltda, Juiz de Fora
  - ICM - Instituto do Coracao de Marilia, Marília
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Monte Alegre
  - Dom Vicente Scherer Hospital, Porto Alegre
  - Hospital de Clínicas de Porto Alegre - Nephrology, Porto Alegre
  - Centro de Pesquisa Clinica Professor Salomao Kelner, Recife
  - Hospital São Lucas, Rio de Janeiro
  - Hospital Universitario Pedro Ernesto - Departamento de Nefrologia, Rio de Janeiro
  - Hospital Universitario Pedro Ernesto - Departamento de Patologia, Rio de Janeiro
  - Comlexo Hospitalar Universitário Professor Edgard Santos, Salvador
  - CSB Group of Nephrology Brazil, Salvador
  - Hospital Ana Nery/SESAB, Salvador
  - Praxis Pesquisa Medica, Santo André
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
  - Hospital das Clínicas da Faculdade de Medicina - Laboratório de Nefrologia Celular, Genética e Molecular, São Paulo
  - Hospital do Rim - Fundação Oswaldo Ramos, São Paulo
  - Hospital Nove de Julho - Nephrology, São Paulo
  - Irmandade Da Santa Casa De Misericordia De Sao Paulo, São Paulo
- Canada (2):
  - Recherche GCP Research, Montreal
  - Women's College Hospital, Toronto
- Colombia (7):
  - Clinica de La Costa S.A.S, Atlántico
  - Solano & Terront Servicios Medicos SAS - Unidad Integral de Endocrinologia - UNIENDO, Bogotá
  - Fundación Valle Del Lili, Cali
  - Centro Cardiovascular Aristides Sotomayor Santa Lucía SAS IPS, Cartagena
  - Mediservis del Tolima IPS S.A.S., Ibagué
  - Fundación Hospitalaria San Vicente de Paul, Medellín
  - Promotora Medica Las Americas S.A. - Clinica Las Americas, Medellín
- France (12):
  - Hopital Henri Mondor - Nephrology, Créteil
  - Hospital Nord Michallon - Nephrology, Grenoble
  - Bicetre Hospital, Le Kremlin-Bicêtre
  - CHU Dupuytren 2 - Néphrologie, dialyse, transplantations, Limoges
  - Hôpital de la Conception, Marseille
  - Ambroise Paré Hospital, Paris
  - Hopital Necker Enfants Malades - Nephrology, Paris
  - Hopital Tenon, Paris
  - Université Paris-Descartes / Hôpital Européen Georges Pompidou, Paris
  - CHU de Guadeloupe, Pointe à Pitre
  - AURA Nord, Saint-Ouen
  - Hopital de Rangueil, Toulouse
- Ghana (3):
  - University of Ghana Medical School - Nephrology, Accra
  - The Bank Hospital, Cantonments
  - Komfo Anokye Teaching Hospital - Nephrology, Kumasi
- Amsterdam UMC - Amsterdam Public Health Research Institute, Amsterdam, Netherlands
- Nigeria (5):
  - University of Nigeria Teaching Hospital, Enugu
  - University College Hospital, Ibadan
  - Lagos University Teaching Hospital, Idi Araba
  - Lagos State University Teaching Hospital, Ikeja
  - Nigerian Institute of Medical Research, Lagos
- Portugal (4):
  - Unidade Local de Saude Amadora/Sintra, E.P.E., Amadora
  - Hospital Curry Cabral - Serviço de Nefrologia, Lisbon
  - Unidade Local de Saúde de Santa Maria, E.P.E. - Nephrology, Lisbon
  - Unidade Local de Saúde de Loures-Odivelas, E.P.E., Loures
- Puerto Rico (3):
  - FDI Clinical Research, Mayagüez
  - University of Puerto Rico, Rio Piedras
  - GCM Medical Group, PSC, San Juan
- Spain (5):
  - Hospital Clinic de Barcelona - Nephrology, Barcelona
  - Hospital Universitari Vall d´Hebron - Servicio de Pediatria, Barcelona
  - Reina Sofia University Hospital - Nephrology, Córdoba
  - Hospital Universitario 12 de Octubre - Nephrology, Madrid
  - Hospital Universitario Virgen Macarena, Seville
- United Kingdom (18):
  - Mid and South Essex Hospitals NHS Trust, Basildon
  - Synexus Clinical Research - Glasgow (DRS), Bellshill
  - FutureMeds Birmingham, Birmingham
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Synexus Clinical Research - Midlands (DRS), Birmingham
  - Epsom and St Helier University Hospitals NHS Trust, Carshalton
  - Leicester General Hospital, Leicester
  - Great Ormond Street Hospital for Children, London
  - Guy's Hospital - Endocrinology, London
  - King's College Hospital - Pulmonology, London
  - Royal Free Hospital - Nephrology, London
  - St George's Hospital London - Nephrology, London
  - St Pancras Clinical Research, London
  - The Royal London Hospital - Nephrology, London
  - Manchester Royal Infirmary - Endocrinology, Manchester
  - Synexus Clinical Research - NW Consortium Manchester (DRS), Manchester
  - Wythenshawe Hospital - Medicines Evaluation Unit, Manchester
  - Nottingham University Hospitals - Children's Clinical Research Facility - Pulmonology, Nottingham

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/